CLINICAL TRIAL: NCT02549976
Title: Evaluation of Digestive Damage and Associated Predictive Factors in Crohn's Disease 5 to 10 Years After Diagnosis
Acronym: DESTIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Groupe d'Etude Therapeutique des Affections Inflammatoires Digestives (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-4
Record Dates: First submitted 2015-09-11; First posted 2015-09-15 (Estimated); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease; Digestive Damage; Lemann Index
MeSH Terms: conditions — Crohn Disease | interventions — Gastroscopy; Colonoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Evaluation group (Experimental): Digestive damage will be assessed on patients by using the methods described in the Lemann index protocol, dependant of Crohn's disease locations.
  All patients will have clinical examination and abdominal magnetic resonance imaging analyses. Upper endoscopy, colonoscopy, and pelvic magnetic resonance imaging analyses will be performed according to disease locations :
  * Upper tract location : upper endoscopy
  * Colorectal location : colonoscopy
  * Perianal location : pelvic MRI
  * All patients : abdominal MRI
  Interventions: Procedure: Abdominal MRI; Procedure: Upper endoscopy; Procedure: Colonoscopy; Procedure: Pelvic MRI

INTERVENTIONS:
Procedure: Abdominal MRI — Abdominal MRI to realize within 4 months following inclusion
Procedure: Upper endoscopy — Upper endoscopy to realize within 4 months following inclusion
Procedure: Colonoscopy — Colonoscopy to realize within 4 months following inclusion
Procedure: Pelvic MRI — Pelvic MRI to realize within 4 months following inclusion

SUMMARY:
The primary objective is to evaluate digestive damage in CD 5 to 10 years after diagnosis in the GETAID centers included in the RAPID study. Secondary objective is to identify predictive factors of the evolution digestive damage.

DETAILED DESCRIPTION:
Background: Crohn's disease (CD) is a chronic inflammatory disorder of the bowel that is characterized by periods of clinical remission alternating with periods of recurrence. Persistent inflammation is believed to lead to progressive bowel damage that, over time, will manifest in the development of strictures, fistulae, and abscesses. The recent development of the Lemann index allows us to precisely assess digestive damage in CD. The aim of the present study is to evaluate digestive damage and associated predictive factors in CD 5 to 10 years after diagnosis.

Methods: Prospective, multicenter, international, transversal, observational study. Patients who completed the RAPID trial (evaluating the benefits on the course of CD of an early prescription of azathioprine compared with conventional step-care therapy) will be eligible. Digestive damage will be assessed using methods described in the Lemann index protocol, dependent on CD location (abdominal MRI obligatory). The total duration of study participation for 1patient will be ≤4 months.

Aims: The primary objective is to evaluate digestive damage in CD 5 to 10 years after diagnosis in the GETAID centers included in the RAPID study. Secondary objective is to identify predictive factors of the evolution digestive damage.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients over 18 years old
* Active or Inactive Crohn's Disease
* Previously enrolled in RAPID clinical trial

Exclusion Criteria:

* Pregnant or nursing woman
* Patient with a contraindication or who decline to have study exams (MRI and endoscopy)
* Other medical or psychiatric or serious chronic conditions or according to the physician's discretion that could affect the patient's cooperation or the capacity to follow study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Digestive damage | 5 to 10 years after diagnosis
  Evaluate digestive damage in Crohn's Disease by using Lemann Index

SECONDARY OUTCOMES:
Predictive factors of the digestive damage evolution | 5 to 10 years after diagnosis
  Evaluate digestive damage per organ (upper intestinal tract, small bowel, colon or rectum, anal or perianal) by using Lemann Index
Predictive factors of the digestive damage evolution | 5 to 10 years after diagnosis
  Determine correlation between Lemann Index and factors measured at diagnosis and then 5 to 10 years after diagnosis.
Variation of Lemann Index | 5 to 10 years after diagnosis
  Variation of Lemann Index 5 to 10 years after diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Pariente, MD, PhD, Principal Investigator — Groupe d'Etude Therapeutique des Affections Inflammatoires Digestives; Jacques Cosnes, MD, Principal Investigator — Groupe d'Etude Therapeutique des Affections Inflammatoires Digestives
Locations (9):
- France (9):
  - Chu Clermont-Ferrand, Clermont-Ferrand
  - Hopital Beaujon, Clichy
  - CHRU Lille, Lille
  - CHU NICE, Nice
  - Hopital Saint Louis, Paris
  - Hopital Saint-Antoine, Paris
  - IMM, Paris
  - CHU Bordeaux - Pessac, Pessac
  - Chu Toulouse, Toulouse

REFERENCES:
- [Background] Pariente B, Mary JY, Danese S, Chowers Y, De Cruz P, D'Haens G, Loftus EV Jr, Louis E, Panes J, Scholmerich J, Schreiber S, Vecchi M, Branche J, Bruining D, Fiorino G, Herzog M, Kamm MA, Klein A, Lewin M, Meunier P, Ordas I, Strauch U, Tontini GE, Zagdanski AM, Bonifacio C, Rimola J, Nachury M, Leroy C, Sandborn W, Colombel JF, Cosnes J. Development of the Lemann index to assess digestive tract damage in patients with Crohn's disease. Gastroenterology. 2015 Jan;148(1):52-63.e3. doi: 10.1053/j.gastro.2014.09.015. Epub 2014 Sep 21. PMID 25241327
- [Background] Cosnes J, Bourrier A, Laharie D, Nahon S, Bouhnik Y, Carbonnel F, Allez M, Dupas JL, Reimund JM, Savoye G, Jouet P, Moreau J, Mary JY, Colombel JF; Groupe d'Etude Therapeutique des Affections Inflammatoires du Tube Digestif (GETAID). Early administration of azathioprine vs conventional management of Crohn's Disease: a randomized controlled trial. Gastroenterology. 2013 Oct;145(4):758-65.e2; quiz e14-5. doi: 10.1053/j.gastro.2013.04.048. Epub 2013 Apr 30. PMID 23644079
- See also: Related Info — http://www.getaid.org